CLINICAL TRIAL: NCT03142945
Title: Mechanical Diagnosis and Therapy vs Traditional Physical Therapy in the Treatment of Mechanical Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Collaborators: Mary Free Bed Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Daniel Vaughn, Professor, Department of Physical Therapy, Grand Valley State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrandVSU
Record Dates: First submitted 2017-04-25; First posted 2017-05-08 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Headaches, Tension
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Intervention Model Description: Two randomized groups. One receiving traditional physical therapy treatments for patients with mechanical headaches. The other will receive an MDT- based approach.
Who Masked: Participant
Masking Description: Patients will not be advised of their group until they exit the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physical Therapy Group (Active Comparator): Traditional Physical Therapy Group Physical therapy-based interventions: home exercises (not repeated motions), stretching, modalities, and posture instruction.
  Interventions: Other: Traditional Physical Therapy
- MDT based physical therapy (Experimental): MDT based physical therapy Physical therapy-based interventions: home exercises (including repeated motions), stretching, modalities, and posture instruction.
  Interventions: Other: MDT based physical therapy

INTERVENTIONS:
Other: Traditional Physical Therapy — Physical therapy-based interventions
  Arms: Traditional Physical Therapy Group
Other: MDT based physical therapy — MDT based physical therapy
  Arms: MDT based physical therapy

SUMMARY:
In addition to manual therapy, mobilizations, manipulations, and exercise, the McKenzie method of Mechanical Diagnosis and Therapy (MDT) is currently being used to treat headaches. However, there is little supportive evidence about the efficacy of this type of treatment. The MDT method focuses on actively involving the patient in education and self-management of pain. The focus is to have the patient learn about his/her condition and how to manage the symptoms independently when possible.

With regards to research that has been conducted on the use of MDT with headaches, one study compared mechanical traction, rhythmic impulse, and MDT exercises in relieving tension-type headaches (TTH). Mechanical cervical traction was found to be more effective at reducing headaches in both infrequent episodic and frequent episodic TTH. While MDT was used in this study, a general treatment was prescribed to each patient in that group without consideration to directional preference. This treatment had the patients perform the same exercises in the same progression, including four extension exercises, one flexion exercise, two lateral flexion exercise, and one rotation exercise. In addition, they performed the exercises for the same length of time for the same number of repetitions. The study was unclear about whether the exercises were administered by physical therapists or whether the practitioners were MDT credentialed.

One case study described the treatment of a cervicogenic headache using the MDT retraction progression along with therapeutic exercises that included deep neck flexor and extensor strengthening and stretching of neck musculature as indicated . The patient reported that performing retractions at home provided him relief from his headaches for progressively longer periods of time as his treatment progressed. By the end of the treatment, the patient no longer experienced headaches. The results from this article support the proposition that headaches which present with mechanical origins can be successfully treated with the MDT approach.

DETAILED DESCRIPTION:
Headaches affect an estimated 46% of adults worldwide, and the pain can have a detrimental effect on an individual's livelihood. In a two-week time period, 12.7% of the US workforce was unable to productively work due to pain, with headache pain as the most common complaint. For those with headache pain, this resulted in 3.5 +/- 0.1 hours of productivity lost in a week. Quality of life, financial situation, employment, and social involvement are negatively impacted by headache pain. Coworkers and family may have to handle work or personal responsibilities that those with headaches are unable to fulfill.

In addition to manual therapy, mobilizations, manipulations, and exercise, the McKenzie method of Mechanical Diagnosis and Therapy (MDT) is currently being used to treat headaches. However, there is little supportive evidence about the efficacy of this type of treatment. The MDT method focuses on actively involving the patient in education and self-management of pain. The focus is to have the patient learn about his/her condition and how to manage the symptoms independently when possible.

A study in Poland compared MDT interventions to a control group that received therapeutic exercise, massage, and ultra-red radiation for patients with cervical derangement. Although not targeted at patients with a primary complaint of headache, the percentage of patients in the MDT group experiencing headache decreased from 80% to 3.33% whereas the percentage of patients in the control group experiencing headaches decreased from 83.87% to 51.61%. This indicates that MDT may be an effective treatment for headaches with a mechanical component.

With regards to research that has been conducted on the use of MDT with headaches, one study compared mechanical traction, rhythmic impulse, and MDT exercises in relieving TTH. Mechanical cervical traction was found to be more effective at reducing headaches in both infrequent episodic and frequent episodic TTH. While MDT was used in this study, a general treatment was prescribed to each patient in that group without consideration to directional preference. This treatment had the patients perform the same exercises in the same progression, including four extension exercises, one flexion exercise, two lateral flexion exercise, and one rotation exercise. In addition, they performed the exercises for the same length of time for the same number of repetitions. The study was unclear about whether the exercises were administered by physical therapists or whether the practitioners were MDT credentialed.

One case study described the treatment of a cervicogenic headache using the MDT retraction progression along with therapeutic exercises that included deep neck flexor and extensor strengthening and stretching of neck musculature as indicated . The patient reported that performing retractions at home provided him relief from his headaches for progressively longer periods of time as his treatment progressed. By the end of the treatment, the patient no longer experienced headaches. The results from this article support the proposition that headaches which present with mechanical origins can be successfully treated with the MDT approach.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old: documentation ie: driver's license
2. Decrease in active cervical range of motion, compared to normal values established by Magee [8]: Measured by Mary Free Bed physical therapists using the Cervical Range of Motion inclinometer (i.e., the CROM).
3. Headache symptoms change based on manual pressure to cervical spine, posture, or neck movement: Tested by Mary Free Bed physical therapist during evaluation
4. Cognition adequate for understanding (alert and oriented x3): Tested by Mary Free Bed physical therapists
5. English-speaking, or able to understand English well enough to follow directions: Determined at initial evaluation. Translators will not be available during the study due to lack of funding and availability.

Exclusion Criteria:

1. Cervical spine fusion less than 6 months: Medical documentation and history portion of initial evaluation. Medical documentation to be reviewed will only be viewed by the physical therapist and will only include information that is typically available to physical therapists in standard practice.
2. Trauma to neck or head within the past 3 months: Medical documentation and history portion of initial evaluation
3. Concussion currently undergoing treatment: Medical documentation and history portion of initial evaluation
4. Signs and symptoms of vertebral artery insufficiency: history portion of initial evaluation and potentially the vertebral artery test performed by the Mary Free Bed physical therapists
5. Diagnosis of Rheumatoid Arthritis or Down Syndrome: Medical documentation and history portion of initial evaluation
6. Constitutional signs or symptoms: nausea, vomiting, profuse sweating, dizziness, etc related to systemic illness: history portion of initial evaluation
7. Signs and symptoms of poor upper cervical spine ligament integrity: Identified through specific manual upper cervical ligament tests performed by the Mary Free Bed physical therapists
8. Connective tissue disorders: Ehlers-Danlos: Medical documentation and history portion of initial evaluation
9. Chiari malformation: Medical documentation and history portion of initial evaluation
10. Signs and symptoms or evidence of myelopathy: Medical documentation and history portion of initial evaluation
11. Diagnosis of dissociative personality disorder: Medical documentation and history portion of initial evaluation
12. Pregnant: Medical documentation and history portion of initial evaluation
13. Neuropsychology issues such as inability to follow multistep directions and short term memory loss: Medical documentation and history portion of initial evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 3 weeks
  functional questionnaire

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 3 weeks
  Pain scale
Cervical Spine Range of Motion | 3 weeks
  Active Range of Motion

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Bacon-Baguley, PhD, Study Chair — Grand Valley State University
Locations (1):
- Grand Valley State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No